CLINICAL TRIAL: NCT02428790
Title: Gastrointestinal Transit Time in Patients With Severe Acquired Brain Injury
Status: Completed | Type: Observational
Sponsor: University of Aarhus (Other)
Collaborators: Aarhus University Hospital (Other); Regionshospitalet Hammel Neurocenter (Other)
Responsible Party: Sponsor
Other Study IDs: ABITransitTimeHammel
Record Dates: First submitted 2015-04-17; First posted 2015-04-29 (Estimated); Last update posted 2015-12-02 (Estimated); Status verified 2015-01

CONDITIONS: Brain Injury; Constipation
MeSH Terms: conditions — Brain Injuries; Constipation

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- ABI Patients: Patients with acquired brain injury.

SUMMARY:
Empirically patients with acquired brain injury (ABI) are often constipated. This is a major clinical issue. Nevertheless, this has only been sparsely studied.

The investigators will measure gastrointestinal transit time (GITT) in 30 patients with ABI, and compare this to healthy controls. Secondly heart rate variability (HRV) is measured in these patients, and associations between HRV and GITT are investigated.

ELIGIBILITY:
Inclusion Criteria:

* ABI:
* Moderate to severe traumatic brain injury (TBI) (Glasgow Coma Scale (GCS) score 3-12 at admission)
* or Stroke
* or Anoxic brain injury
* Ability to swallow the capsules used to assess GITT
* Ability to give meaningful informed consent to participate in the study

Exclusion Criteria:

* Major abdominal disorders
* Severe acute comorbidity
* Known cancer
* Pregnancy
* Known autonomic neuropathy
* Other known neurological disorder

Ages: 18 Years to 79 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients at Hammel Neurocenter and University Clinic, during rehabilitation after aquired brain injury
Sampling Method: Non-Probability Sample
Enrollment: 25 (Actual)
Dates: Start 2015-05; Primary Completion 2015-11 (Actual); Study Completion 2015-11 (Actual)

PRIMARY OUTCOMES:
Gastrointestinal transit time (GITT) [in days] | During rehabilitation, when the patient meet the inclusion criteria. This is expected to be between 2 weeks and 4 months after the primary injury.

SECONDARY OUTCOMES:
Association between heart rate variability (HRV) and GITT | During rehabilitation, when the patient meet the inclusion criteria. This is expected to be between 2 weeks and 4 months after the primary injury.
  Linear regression with GITT as dependent variable, and high frequency power sepectral density analysis of the heart rate (HF) as the independent variable.

CONTACTS AND LOCATIONS:
Overall Officials: Henning Andersen, Professor, Dr. med. PhD, Principal Investigator — Aarhus University Hospital